CLINICAL TRIAL: NCT00886184
Title: Intra-arrest Therapeutic Hypothermia in Prehospital Cardiac Arrest. Impact on Biomarker of Brain Damage.
Brief Title: Intra-arrest Therapeutic Hypothermia in Prehospital Cardiac Arrest
Acronym: HITUPPAC-BIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0821; 2008-A01488-47 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2013-01-30 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Arrest
Keywords: Hypothermia; Cardiac arrest; Biomarkers; Pre hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Induction of pre hospital early hypothermia in patients having a cardiac .
  Interventions: Procedure: Hypothermia.
- 2 (Active Comparator): Induction of hypothermia only at hospital arrival.
  Interventions: Procedure: No early hypothermia

INTERVENTIONS:
Procedure: Hypothermia. — Induction of pre hospital therapeutic hypothermia.
  Arms: 1
Procedure: No early hypothermia — Induction of therapeutic hypothermia only once arrived at hospital.
  Arms: 2

SUMMARY:
The aim is to precise the place of therapeutic hypothermia induced before Return of Spontaneous Circulation (ROSC) in pre hospital cardiac arrest. If we find a benefit in terms of biomarkers in inducing in early hypothermia compared to hypothermia induced only after arrival at the hospital, there will be arguments to develop a higher scale study, allowing to prove benefits in terms of survival and neurological status.

DETAILED DESCRIPTION:
Principal aim : prove the efficiency of early therapeutic hypothermia induced during ischemia in pre hospital cardiac arrest by a reduction of brain damage biomarkers.

Secondary aim: prove the efficiency of early therapeutic induced hypothermia in the reduction of pro-inflammatory cytokines secretion. Determine the number of ROSC, patients survival, neurological status 48 hours after cardiac arrest (GCS) and when leaving the hospital, impact following initial cardiac rhythm and the cooling rate of early therapeutic induced hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* pre hospital cardiac arrest

Exclusion Criteria:

* under 18 years old
* pregnancy or breastfeeding women
* patient under guardianship.
* not beneficing a social health care system.
* cardiac arrest of traumatic origin
* patients with an initial body temperature under 34° C
* cardiac arrests for which resuscitation maneuvers seem unjustified (DNR criteria)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2009-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Prove efficacy of early induced hypothermia during ischemia in pre hospital cardiac arrest by a reduction of brain damage biomarkers. | 72 hours

SECONDARY OUTCOMES:
Prove the efficacy of early therapeutic induced hypothermia in the reduction of pro-inflammatory cytokines secretion. | 72 hours
Determine the number of Return of Spontaneous Circulation (ROSC), patients survival. | 72 hours
Determine neurological status 48 hours after cardiac arrest (GCS) | 48 hours
Determine impact following initial cardiac rhythm. | 72 hours
Determine the cooling rate of early therapeutic induced hypothermia. | 72 hours
Determine neurological status when leaving hospital (or 28 days if not applicable) (CPC) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DEBATY, MD, Principal Investigator — Emergency department - Mobile Intensive Care Unit
Locations (1):
- University Hospital Grenoble, Grenoble, France

REFERENCES:
- [Derived] Ferreira Da Silva IR, Frontera JA. Targeted temperature management in survivors of cardiac arrest. Cardiol Clin. 2013 Nov;31(4):637-55, ix. doi: 10.1016/j.ccl.2013.07.010. PMID 24188226